CLINICAL TRIAL: NCT02269280
Title: Phase II Randomized Study of Lower Doses of Decitabine (DAC; 20 mg/m2 IV Daily for 3 Days Every Month) Versus Azacitidine (AZA; 75 mg/m2 SC/IV Daily for 3 Days Every Month) Versus Azacitidine (AZA; 75 mg/m2 SC/IV Daily for 5 Days Every Month) in MDS Patients With Low and Intermediate-1 Risk Disease Transfusion-Dependent Versus Best Supportive Care (BSC) in MDS Patients With Low and Intermediate-1 Risk Disease Transfusion-Independent
Brief Title: Phase II Decitabine (DAC) Versus Azacitidine (AZA) in Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0112; NCI-2014-02339 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0112 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-10-13; First posted 2014-10-21 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic syndrome; MDS; Low or intermediate-1 risk; Transfusion-dependent; Transfusion-independent; Best supportive care; BSC; Azacitidine; 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine; Decitabine; Dacogen
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Azacitidine (AZA) - Days 1 - 3 (Experimental): Azacitidine (AZA) Azacitidine 75 mg/m2 by vein or subcutaneously daily for 3 days (days 1-3) approximately every 28 days.
  Interventions: Drug: Azacitidine (AZA) Days 1 - 3
- Azacitidine (AZA) - Days 1 - 5 (Experimental): Azacitidine (AZA) 75 mg/m2 by vein or subcutaneously daily for 5 days (days 1-5) approximately every 28 days.
  Interventions: Drug: Azacitidine (AZA) Days 1 - 5
- Decitabine (DAC) (Experimental): Decitabine 20 mg/m2 by vein for 3 days (days 1-3) approximately every 28 days.
  Interventions: Drug: Decitabine (DAC)
- Best Supportive Care (BSC) (Other): Participants receive standard of care as chosen by study doctor. Best supportive care for transfusion-independent participants only.
  Interventions: Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Azacitidine (AZA) Days 1 - 3 — Azacitidine 75 mg/m2 by vein or subcutaneously daily for 3 days (days 1-3) approximately every 28 days.
  Other Names: 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
  Arms: Azacitidine (AZA) - Days 1 - 3
Drug: Decitabine (DAC) — Decitabine 20 mg/m2 by vein for 3 days (days 1-3) approximately every 28 days.
  Other Names: Dacogen
  Arms: Decitabine (DAC)
Other: Best Supportive Care (BSC) — Participants receive standard of care as chosen by study doctor. Best supportive care for transfusion-independent participants only.
  Arms: Best Supportive Care (BSC)
Drug: Azacitidine (AZA) Days 1 - 5 — Azacitidine 75 mg/m2 by vein or subcutaneously daily for 5 days (days 1-5) approximately every 28 days.
  Other Names: 5-Azacytidine; 5-AZA; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
  Arms: Azacitidine (AZA) - Days 1 - 5

SUMMARY:
The goal of this clinical research study is to compare how 2 different drugs, decitabine and azacitidine, when given on a shorter than standard dosing schedule, may help to control MDS. The safety of each study drug given on these schedules will also be studied.

This is an investigational study. Decitabine and azacitidine are both FDA approved and commercially available for use in patients with MDS. Giving these drugs on a different schedule than is standard is considered investigational.

The study doctor can tell you how the study drugs are designed to work.

DETAILED DESCRIPTION:
Study Groups and Study Drug Administration:

Each cycle is approximately 28 days.

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to 1 of 4 groups:

* If you are in Group 1, you will receive decitabine by vein over about 1 hour on Days 1-3 of every cycle.
* If you are in Group 2, you will receive azacitidine either as an injection under your skin or by vein on Days 1-3 of every cycle.
* If you are in Group 3, you will receive azacitidine either as an injection under your skin or by vein on Days 1-5 of every cycle.
* If you are in Group 4, you will receive the standard of care. The study doctor can explain the treatment you will receive and the risks involved.

Transfusion-dependent participants will be randomly assigned to 1 of 3 groups

This is done because no one knows if one study group is better, the same, or worse than the other group. If you are among the first 20 participants, you will have an equal chance of being in any of the groups. If you enroll after that, you will have a higher chance of being assigned to the group that has had better results.

However, once you are assigned to a group, you will not be allowed to change groups.

You may be given other drugs to help prevent side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Study Visits:

One (1) time each month, blood (about 2 tablespoons) will be drawn for routine tests.

At the end of Cycle 2, then every 3 cycles for the first year, then every 6 cycles, you will have a bone marrow biopsy and/or aspirate to check the status of the disease and for cytogenetic testing.

After Cycle 1, if the study doctor decides it is acceptable, you may be allowed to receive treatment from your local cancer doctor. However, you must return to Houston at least every 3 cycles for study visits. How often these visits will occur will depend on what the doctor thinks is in your best interest.

Length of Study:

You may continue taking the study drug or standard therapy for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug or standard therapy if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Follow-Up:

When you are off-treatment, every 6 -12 months for up to 5 years, you will be called by a member of the study staff. You will be asked about any side effects you may be having. The phone calls will take about 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an IRB-approved informed consent document.
2. Age >/= 18 years.
3. IPSS low- or intermediate-1-risk MDS, including CMML-1
4. ECOG performance status of </= 3 at study entry.
5. Organ function defined as: Serum creatinine </= 2 mg/dL; Total bilirubin </= 2 x ULN; ALT (SGPT) </= 2 x ULN; AST (SGOT) </= 2 x ULN
6. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days and will also need to use contraceptives. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential.

Exclusion Criteria:

1. Breast feeding females
2. Prior therapy with decitabine or azacitidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, Principal Investigator — M.D. Anderson Cancer Center
Locations (6):
- United States (6):
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NYP/Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azacitidine (AZA) - Days 1 - 3 | Azacitidine (AZA) - Days 1 - 5 | Decitabine (DAC) | Best Supportive Care (BSC)
Started | 54 | 68 | 58 | 5
Completed | 54 | 68 | 58 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azacitidine (AZA) - Days 1 - 3 | Azacitidine (AZA) - Days 1 - 5 | Decitabine (DAC) | Best Supportive Care (BSC) | Total
Number analyzed (Participants) | 54 | 68 | 58 | 5 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 14 | 2 | 51
  >=65 years | 38 | 49 | 44 | 3 | 134
Age, Continuous [Median (Full Range); unit: years] | 72 [24 to 85] | 70 [29 to 85] | 71 [55 to 85] | 67 [61 to 74] | 71 [24 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 16 | 1 | 47
  Male | 41 | 51 | 42 | 4 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 5 | 0 | 7
  White | 50 | 65 | 48 | 5 | 168
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 54 | 68 | 58 | 5 | 185

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival (EFS)
Description: Event free survival (EFS) defined as the time from beginning of treatment till an event occurs or last follow-up. For transfusion independent patients, the events includes lack of response, requirement of blood transfusion, progression to advanced stages of disease, transformation into AML, discontinuation of therapy due to side effects, and death.
  For transfusion dependent patients, the events includes lack of response, progression to advanced stages of disease, transformation into AML, discontinuation of therapy due to side effects, and death.
Time Frame: Up to 8 years, 9 months and 12 days
Measure: Median (Full Range); unit: Months
Arm/Group | Azacitidine (AZA) - Days 1 - 3 | Azacitidine (AZA) - Days 1 - 5 | Decitabine (DAC) | Best Supportive Care (BSC)
Number analyzed (Participants) | 54 | 68 | 58 | 5
Months | 14.1 [1.1 to 75.4] | 18.0 [0.9 to 61.6] | 9.8 [0.8 to 31.0] | 13.3 [0.8 to 75.4]

2. Secondary Outcome: Number of Participants With Overall Improvement
Description: Overall improvement, defined as complete remission (CR), partial remission (PR), marrow CR (mCR), or hematologic improvement (HI), measured using each patient's best response with the 2 different agents. Response assessed using the modified MDS International Working Group 2006 criteria.
Time Frame: Up to 8 years, 9 months and 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Azacitidine (AZA) - Days 1 - 3 | Azacitidine (AZA) - Days 1 - 5 | Decitabine (DAC) | Best Supportive Care (BSC)
Number analyzed (Participants) | 54 | 68 | 58 | 5
Participants | 22 | 27 | 29 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 years, 9 months and 12 days
Arm/Group | Azacitidine (AZA) - Days 1 - 3 | Azacitidine (AZA) - Days 1 - 5 | Decitabine (DAC) | Best Supportive Care (BSC)
All-Cause Mortality (participants affected / at risk) | 1/54 | 2/68 | 5/58 | 0/5
Serious Adverse Events (participants affected / at risk) | 4/54 | 3/68 | 0/58 | 0/5
Other Adverse Events (participants affected / at risk) | 35/54 | 51/68 | 38/58 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (AZA) - Days 1 - 3 (N=54) | Azacitidine (AZA) - Days 1 - 5 (N=68) | Decitabine (DAC) (N=58) | Best Supportive Care (BSC) (N=5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (AZA) - Days 1 - 3 (N=54) | Azacitidine (AZA) - Days 1 - 5 (N=68) | Decitabine (DAC) (N=58) | Best Supportive Care (BSC) (N=5)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 3 (3) | 3 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (10) | 3 (3) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 9 (13) | 2 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 3 (3) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 3 (7) | 1 (2) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (6) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 3 (3) | 7 (8) | 1 (8) | 1 (1)
Fatigue (General disorders) | 2 (2) | 9 (11) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 5 (5) | 5 (8) | 0 (0)
Fever (General disorders) | 3 (3) | 4 (5) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (6) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 4 (7) | 1 (1) | 6 (6) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5) | 5 (6) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 5 (5) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 10 (63) | 24 (81) | 13 (59) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Platelet count decreased (Infections and infestations) | 3 (13) | 13 (41) | 14 (62) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (6) | 5 (9) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 4 (8) | 2 (3) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 2 (4) | 6 (21) | 4 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT02269280/Prot_SAP_000.pdf